CLINICAL TRIAL: NCT05299034
Title: Treatment of Stroke in the Extended Window: Optimization of the Radiological Selection and Transfer Model in Patients With a Stroke Presenting 6-24h After Symptoms Onset (VESTA Study)
Brief Title: Optimizing the Radiological Selection and Transfer Model in Stroke Patients Presenting 6-24h After Onset (VESTA Study)
Acronym: VESTA
Status: Completed | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, María Hernández Pérez, MD, PhD, Germans Trias i Pujol Hospital
Other Study IDs: PI21/01548
Record Dates: First submitted 2022-01-13; First posted 2022-03-28 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients 6-24h receiving non-contrast CT + CTA: Stroke patients 6-24h undergoing non-contrast CT + CTA to decide stroke therapy
  Interventions: Diagnostic Test: Non contrast CT+CT angiography
- Stroke patients 6-24h receiving multimodal imaging: Stroke patients 6-24h undergoing NCCT+CTA+CTP or MRI with DWI and PWI imaging to decide stroke therapy
  Interventions: Diagnostic Test: Multiparametric imaging

INTERVENTIONS:
Diagnostic Test: Multiparametric imaging — MR perfusion or multiparametric CT including NCCT, CTA and CTP
  Groups: Stroke patients 6-24h receiving multimodal imaging
Diagnostic Test: Non contrast CT+CT angiography — NCCT+CTA
  Groups: Stroke patients 6-24h receiving non-contrast CT + CTA

SUMMARY:
We aim to optimize the radiological selection and the transfer model in patients with a 6-24h stroke for a fairer and broader access to a reperfusion treatment. The specific objectives are:

1. To confirm that the selection of patients for reperfusion therapies in the late window is safe by applying the same clinical and imaging criteria recommended by clinical guidelines for the early window treatment selection.
2. To evaluate the performance of non-contrast CT by applying immediate post-processing software for the selection of patients for reperfusion treatment in the late window.
3. To analyze the prehospital and arrival variables at the primary stroke center to generate decision trees that optimize the transfer decision in patients with activation of the stroke code in >6h from the onset of symptoms.

METHODOLOGY: Study based on a mandatory, prospective, multicenter registry (CICAT registry) consisting of two phases

1. retrospective analysis with a detailed evaluation of the images of the included patients and generation of "machine learning" models that accurately predict the probability of receiving reperfusion treatment in the late window.
2. validation of the models in a prospective study. Clinical, radiological and transport variables will be studied.

Response variables: rate of patients receiving reperfusion treatment in the late window, functional prognosis at 90 days, hemorrhagic transformation, and mortality.

ELIGIBILITY:
* SUBSTUDY 1. OPTIMIZATION OF IMAGING SELECTION METHODS FOR SELECTING STROKE PATIENTS FOR REPERFUSION TREATMENT IN THE EXTENDED WINDOW.

  - Inclusion criteria: Consecutive patients registered in the CICAT registry between the years 2019 and 2021 with a stroke who meet the following criteria
  1. Age older than 18 years,
  2. Diagnosis of acute cerebral infarction,
  3. More than six hours of evolution or uncertain chronology of symptoms,
  4. Absence of disability prior to stroke (modified Rankin score 0-2),
  5. NIHSS score>5,
  6. Neuroimaging study including at least one non-contrast cranial CT scan within 60 minutes of arrival at the hospital center.
* SUBSTUDY 2. OPTIMIZATION OF CIRCUITS AND TRANSFER MODEL IN PATIENTS WITH STROKE IN THE EXTENDED WINDOW OF TREATMENT.

  * Inclusion criteria: Selection of consecutive, prospective patients to be included in the CICAT registry between January 2023 and March 2024 with stroke meeting the following criteria:

    1. Age over 18 years,
    2. Suspicion of acute cerebral infarction,
    3. More than six hours of evolution or uncertain chronology of symptoms,
    4. absence of pre-stroke disability (modified Rankin score 0-2),
    5. NIHSS score greater than 5.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with stroke suspiction in Catalonia included in the CICAT registry
Sampling Method: Non-Probability Sample
Enrollment: 2173 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
mRS at 90 days | 90 days after stroke
  Percentage of patients with functional independence, defined as mRS < or =2 on day 90 as assessed centrally by blinded evaluators of the Catalan Stroke Master Plan.
Rate of patients treated with mechanical thrombectomy | less than 24 hours after the diagnostic test

SECONDARY OUTCOMES:
Mortality at discharge and at day 90 | 90 days after stroke
Symptomatic intracerebral hemorrhage, defined as PH2 or SAH on imaging test at 24-72 hours associated with a worsening in NIHSS ≥ 4 points | From 24 to 72 hours after stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain